CLINICAL TRIAL: NCT02737059
Title: A Phase I Randomized, Double-Blinded, Placebo-Controlled Study of the Effect of Naloxegol on Gastric, Small Bowel, and Colonic Transit in Healthy Subjects
Brief Title: Effect of Naloxegol on Gastric, Small Bowel, and Colonic Transit in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michael Camilleri (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Michael Camilleri, MD, Consultant, Professor of Medicine, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-007863; UL1TR000135 (NIH)
Record Dates: First submitted 2016-04-08; First posted 2016-04-13 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Constipation Drug Induced
MeSH Terms: interventions — naloxegol; Codeine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Codeine/naloxegol placebo (Placebo Comparator): Each subject will receive two medications to which they are randomized for 1 day before and for the 2 days during transit measurement.
  Codeine tablet 30 mg q.i.d., and placebo tablet matching naloxegol q.d.
  Interventions: Drug: Codeine; Drug: naloxegol placebo
- Naloxegol/ codeine placebo (Placebo Comparator): Each subject will receive two medications to which they are randomized for 1 day before and for the 2 days during transit measurement.
  Naloxegol tablet 25 mg q.d and placebo tablet matching codeine q.i.d.
  Interventions: Drug: Naloxegol; Drug: codeine placebo
- Codeine/ naloxegol (Active Comparator): Each subject will receive two medications to which they are randomized for 1 day before and for the 2 days during transit measurement.
  Codeine tablet 30 mg q.i.d., and naloxegol tablet 25 mg q.d.
  Interventions: Drug: Naloxegol; Drug: Codeine
- codeine placebo/ naloxegol placebo (Active Comparator): Each subject will receive two medications to which they are randomized for 1 day before and for the 2 days during transit measurement.
  Placebo tablet matching codeine q.i.d., and placebo tablet matching naloxegol q.d.
  Interventions: Drug: codeine placebo; Drug: naloxegol placebo

INTERVENTIONS:
Drug: Naloxegol — 25mg daily
  Other Names: MOVANTIK
  Arms: Codeine/ naloxegol; Naloxegol/ codeine placebo
Drug: Codeine — 30mg 4 times daily
  Arms: Codeine/ naloxegol; Codeine/naloxegol placebo
Drug: codeine placebo — 4 times daily (placebo will be made to match the codeine)
  Arms: Naloxegol/ codeine placebo; codeine placebo/ naloxegol placebo
Drug: naloxegol placebo — placebo will match naloxegol, given daily
  Arms: Codeine/naloxegol placebo; codeine placebo/ naloxegol placebo

SUMMARY:
This research study was being done to study the effect of codeine and Naloxegol for 3 days compared to placebo on the movement of food through the colon of healthy individuals. Codeine is a commonly used pain-relieving drug that often causes constipation as an unwanted side effect. Naloxegol is a medication recently approved by the FDA for treatment of constipation induced by Codeine.

The hypothesis for this study was that Naloxegol reduces the retardation of small bowel and colonic transit induced by codeine in healthy participants.

DETAILED DESCRIPTION:
This was a single center, randomized, double-blind, placebo-controlled, parallel-group, Phase I study of the effects of naloxegol, a novel mu-opioid antagonist, on gastrointestinal and colonic transit in the presence or absence of the mu-opiate, codeine. There is a need to develop effective medications for the treatment of opiate-induced constipation and other motility disorders. Currently available opiates are complicated by addictive potential and induction of troublesome constipation.

ELIGIBILITY:
Inclusion criteria:

* Body Mass Index (BMI) between 19 and 30 kg/m^2 and absolute weight between 45 and 100 kg. for both males and females.
* Females who are non-pregnant, non-lactating, postmenopausal for at least one year (as evidenced by last menses 12 months from Day 0), surgically sterile, or willing to use a clinically-approved method of contraception from 35 days prior to Day 0 until 30 days after the last dose of study medication
* Males who are surgically sterile or willing to use a clinically approved method of contraception from Day 0 until 30 days after the last dose of study medication.
* Absence of gastrointestinal symptoms unless deemed not clinically significant by the Investigator.
* Able to understand and willing to sign informed consent
* Negative urine drug screen at screening

Exclusion criteria:

* Structural or metabolic diseases/conditions that affect the gastrointestinal system, or functional gastrointestinal disorders. For screening, three or more "YES" responses on the Bowel Disease Questionnaire will be used to exclude subjects with irritable bowel syndrome.
* Use of drugs or agents within the past 2 weeks or planned use in the subsequent 4 weeks during the study period that: Alter GI transit including laxatives, magnesium or aluminum-containing antacids, prokinetic, erythromycin, narcotics, anticholinergics, tricyclic antidepressants, Selective serotonin re-uptake inhibitors (SSRI) and newer antidepressants.
* Analgesic drugs including opiates, NSAID, cyclooxygenase-2 (COX 2) inhibitors
* Use of non-prescription or prescription medications within 7 days or within five half-lives prior to Day 0 for that particular medication. Note: Low stable doses of thyroid replacement, estrogen replacement, and birth control pills or depot injections, and use of acetaminophen on as needed basis are permissible.
* A score of greater than or equal to 11 for either score obtained from the Hospital Anxiety Depression Scale
* Positive urine drug screen at screening
* Female subjects who are pregnant or breast feeding.
* Clinical evidence (including physical exam, previous laboratory tests) or significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological, psychiatric, or other disease that interfere with the objectives of the study. Patients with previously high transaminase levels (AST, ALT) may be retested and if the results are less than 1.5 times the upper limit of normal will be included as long as they do not have an underlying known liver disease.
* Symptoms of a significant clinical illness in the preceding two weeks.
* Participation in another clinical study within the past 30 days.
* Subjects known allergy or hypersensitive to multiple drug compounds (greater than or equal to 3 drug compounds), naloxegol or opioid antagonists, codeine sulfate, eggs or any components of the study medication
* Daily use of any tobacco products within 6 months prior to Day 0
* Previous exposure to naloxegol
* Any other conditions or prior therapy which, in the opinion of the Investigator, would make the subject unsuitable for this study
* Contraindications to use of naloxegol in accordance with FDA guidance: suspected GI obstruction or at increased risk of recurrent obstruction; concomitant use of strong CYP3A4 inhibitors such as clarithromycin and ketoconazole
* Concomitant treatment with moderate CYP3A4 inhibitors (diltiazem, erythromycin, verapamil) or strong CYP3A4 inducers (rifampin) or other opioid antagonists.
* History of substance abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
Gastric emptying (t1/2) | Day 2
  The time for half of the ingested solids or liquids to leave the stomach.
Colonic filling (%) at 6 hours | Day 2 (6 hours)
  Percent of the radio-labeled meal that reached the colon at 6 hours, indirectly reflecting small bowel transit time.
Colonic geometric center (GC) at 24 hours | Day 2 ( 24 hours)
  The scintigraphic method is used to measure colonic transit. An isotope is adsorbed on activated charcoal particles and delivered to the colon in a delayed release capsule. Anterior and posterior gamma images are taken hourly. The geometric center (GC) is the weighted average of counts in the different colonic regions. The scale ranges from 1 to 5; a high GC implies faster colonic transit, a GC of 1 implies all isotope is in the ascending colon, and a GC of 5 implies all isotope is in the stool.

SECONDARY OUTCOMES:
Colonic transit summarized by GC at 48 hours hours hours colonic transit summarized by GC at 4 and 48 hours Colonic transit at 4 and 48 hours | Day 2 (48 hours)
  The scintigraphic method is used to measure colonic transit. An isotope is adsorbed on activated charcoal particles and delivered to the colon in a delayed release capsule. Anterior and posterior gamma images are taken hourly. The geometric center (GC) is the weighted average of counts in the different colonic regions. The scale ranges from 1 to 5; a high GC implies faster colonic transit, a GC of 1 implies all isotope is in the ascending colon, and a GC of 5 implies all isotope is in the stool.
Ascending Colon Emptying (ACE) T1/2 | Day 2
  Ascending colon emptying half-time will be estimated by power exponential analysis of the proportionate emptying over time of counts from the colon.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No